CLINICAL TRIAL: NCT01635127
Title: A Phase II Randomized Double-Blind Placebo Controlled Single Center Study of Canakinumab Treatment of Adult Patients With Moderate to Severe Chronic Idiopathic Urticaria
Brief Title: Efficacy Study of Canakinumab to Treat Urticaria
Acronym: URTICANA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USZ-DER-AAN-017
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Canakinumab (Experimental): Monoclonal antibody inhibiting interleukin 1 beta
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Constituent, inactive
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — 150mg s.c.
  Other Names: Ilaris
  Arms: Canakinumab
Drug: Placebo — Constituent of canakinumab
  Arms: Placebo

SUMMARY:
Evaluation whether canakinumab leads to improvement of urticaria

DETAILED DESCRIPTION:
Single center prospective placebo-controlled cross-over phase II study.

* To assess if canakinumab can induce clinical improvement and/or complete clinical remission of chronic idiopathic urticaria at week 4 as compared to placebo
* To compare canakinumab and placebo treated patients in the percentage who achieve complete clinical remission at week 1, 2, 4, and 8.
* To compare the percentage with clinical improvement as measured by UAS7 score at week 1, 2, 4, and 8 in canakinumab and placebo treated patients
* To compare the percentage of canakinumab and placebo treated patients with 75% and 100% improvement of their baseline (Run-in-period) UAS7 score at week 1,2,4,and 8
* To compare the daily wheal score for Days 1 to 7 in canakinumab and placebo treated patients

ELIGIBILITY:
Inclusion criteria

* Diagnosis of chronic idiopathic urticaria for more than 6 weeks as confirmed by clinical and, if necessary, histological examination
* CIU of moderate to severe severity defined by all of the following

  * Physician severity score of 2 or 3 (on a scale from 0 - 3)
  * Run-in period of the diary-based UAS7 score of > 21 (on a scale from 0 - 42)
  * Symptomatic despite use of non-sedating antihistamine with or without concomitant leukotriene antagonist/corticosteroids
* Use of maintenance non-sedating antihistamine at a stable dose for at least 1 week prior to entering run-in period
* Maintenance corticosteroids at a dose of <20 mg/day or <0.4 mg/kg stable for at least the week prior to study entry for treatment of the patient's CIU will be allowed.
* Age: > 18 years.
* Signed informed consent
* Negative or unreactive QuantiFERON test (QFT-TB G In-Tube) or history of adequate treatment of active or latent tuberculosis.

Exclusion criteria:

* Age < 18 or > 70 years
* History of cancer except for treated basal cell carcinoma of the skin
* With active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection, active or untreated latent tuberculosis.
* Patients currently treated with systemic immunosuppressive agents or following treatments in the specified period before the baseline visit:

  * corticosteroids =20 mg/day or >0.4 mg/kg for 1 week prior to study entry;
  * leukotriene antagonists for 1 week prior to study entry
  * colchicine, dapsone or mycophenolate mofetil for 3 weeks;
  * etanercept, leflunomide (documentation of a completion of a full cholestyramine elimination treatment after most recent leflunomide use will be required), thalidomide or ciclosporin for 4 weeks;
  * adalimumab or intravenous immunoglobulin for 8 weeks;
  * infliximab, 6-mercaptopurine, azathioprine, cyclophosphamide or chlorambucil for 12 weeks
* Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Pregnant or lactating women, patients (men or women) planning a pregnancy during the duration of the study, lack of safe contraception.
* Safe contraception is defined as follows:
* Double-barrier contraception such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices together with condom use.
* Both men and women must use safe contraception (double-barrier as defined above) during the duration of the study and until 6 months after the study.
* Please note that female subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the subject.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Complete clinical remission | 4 weeks
  Improvement of urticaria within 4 weeks, objective measurements daily wheal score and UAS7

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid-Grendelmeier, Prof MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Switzerland

REFERENCES:
- [Derived] Maul JT, Distler M, Kolios A, Maul LV, Guillet C, Graf N, Imhof L, Lang C, Navarini AA, Schmid-Grendelmeier P. Canakinumab Lacks Efficacy in Treating Adult Patients with Moderate to Severe Chronic Spontaneous Urticaria in a Phase II Randomized Double-Blind Placebo-Controlled Single-Center Study. J Allergy Clin Immunol Pract. 2021 Jan;9(1):463-468.e3. doi: 10.1016/j.jaip.2020.07.058. Epub 2020 Aug 20. PMID 32827729